CLINICAL TRIAL: NCT02320370
Title: Optimizing Electrical Stimulation for Clinical Applications (the OptES Study): Severe Psychological Stress - a Pilot Study (OptES-Stress-pilot)
Brief Title: Transcranial Electrical Stimulation in the Treatment of Acute Anxiety Induced by Stressful Life Events: A Pilot Study
Acronym: OptesStressP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Soili Lehto, Adjunct professor, University of Eastern Finland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OptES-Stress-pilot
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment 1 (Experimental): NeuroConn DC Stimulator Plus tDCS treatment protocol no 1
  Interventions: Device: NeuroConn DC Stimulator Plus tDCS
- Treatment 2 (Experimental): NeuroConn DC Stimulator Plus tDCS treatment protocol no 1
  Interventions: Device: NeuroConn DC Stimulator Plus tDCS

INTERVENTIONS:
Device: NeuroConn DC Stimulator Plus tDCS — transcranial electrical stimulation intervention with two experimental protocols

SUMMARY:
The investigators examine the efficacy of two different transcranial direct current stimulation (tDCS) stimulation protocols in the treatment of acute anxiety in an open-label pilot study in patients who have faced severely stressful life events.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) is a novel neuromodulation method that has been observed to be promising in treatment of psychiatric disorders such as depression. Nevertheless, knowledge related to the treatment of psychological stress and its main symptom, anxiety, is very scarce. The investigators examine the efficacy of two different transcranial direct current stimulation (tDCS) stimulation protocols in the treatment of acute anxiety in an open-label pilot study in patients who have faced severely stressful life events.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Naïve to tDCS
* Right-handed
* Impact of Event Scale Scores ≥ 30

Exclusion Criteria:

* Metal implants inside skull or eye
* Severe skin lesions at the electrode placement area
* History of epilepsy or previous seizures
* Pregnant or breast-feeding
* Pacemaker
* History of intracerebral bleeding during the past six months
* Major psychiatric conditions according to the Structured Clinical Interview for DSM-IV Disorders, i.e., Lifetime diagnoses of bipolar mood disorder or psychotic disorder
* DSM-IV diagnosis for one or more of the following conditions during the past six months: unipolar mood disorder, anxiety disorders, eating disorders, or substance dependence/abuse.
* Use of psychotropic medication (i.e., antipsychotic and antidepressant medications, mood stabilizers, psychostimulants, hypnotics and tranquilizers) during the past six months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Impact of Event Scale (Change in scores of event-related anxiety) | 12 days
  Change in scores of event-related anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Soili M Lehto, MD, PhD, Principal Investigator — University of Eastern Finland